CLINICAL TRIAL: NCT04127721
Title: Itacitinib to Prevent Graft Versus Host Disease
Brief Title: Itacitinib for the Prevention of Graft Versus Host Disease in Patients Undergoing Donor Stem Cell Transplantation
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: 0 ACTUAL Enrollment must have Overall Recruitment Status
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018-0505; NCI-2019-05753 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0505 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-09-30; First posted 2019-10-16 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Allogeneic Stem Cell Transplant Recipient; Hematologic and Lymphocytic Disorder; Hematopoietic and Lymphoid Cell Neoplasm
MeSH Terms: conditions — Hematologic Diseases; Hematologic Neoplasms | interventions — Busulfan; fludarabine; itacitinib; INCB039110; Methotrexate; merphos; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prevention (itacitinib, busulfan, fludarabine, ASCT) (Experimental): CONDITIONING CHEMOTHERAPY: Patients receive busulfan IV over 3 hours on days -20, -13, and -6 to -3, and fludarabine IV over 1 hour on days -6 to -3 in the absence of disease progression or unacceptable toxicity.
  ALLOGENEIC STEM CELL TRANSPLANTATION: Patients undergo ASCT on day 0.
  GVHD PROPHYLAXIS: Patients receive itacitinib PO QD on days -21 to 80. Patients with no evidence of GVHD at day 80 receive a tapered dose of itacitinib until day 90. Patients also receive tacrolimus IV then PO BID for 3 months when able, and methotrexate IV over 30 minutes on days 1, 3, and 6 (day 11 also for patients with a matched unrelated donor).
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Busulfan; Drug: Fludarabine; Drug: Itacitinib; Drug: Methotrexate; Drug: Tacrolimus

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo ASCT
  Other Names: Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT
Drug: Busulfan — Given IV
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Drug: Itacitinib — Given PO
  Other Names: INCB 039110; INCB-039110; INCB039110
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Tacrolimus — Given IV and PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic

SUMMARY:
This phase II trial studies how well itacitinib works in preventing graft versus host disease in patients with blood disorders undergoing donor stem cell transplantation. A donor transplantation uses blood-making cells from a family member or unrelated donor to remove and replace abnormal blood cells. Graft versus host disease is a reaction of the donor's immune cells against the patient's body. Itacitinib plus standard treatment may help prevent graft versus host disease in patients who have received a donor stem cell transplantation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the graft-versus (vs.) host disease-free/relapse free survival (GRFS) rate of itacitinib used as prophylaxis to prevent graft versus host disease (GVHD) after allogeneic stem cell transplantation (ASCT) at one year.

SECONDARY OBJECTIVES:

I. To assess the time to neutrophil and platelet engraftment and compare between matched and unmatched donors.

II. To assess safety of itacitinib as measured by non-relapse mortality (NRM) at day 100.

III. To assess the toxicity profile associated with this regimen. IV. To assess the incidence of acute and chronic GVHD. V. To assess the incidence of disease relapse. VI. To assess the incidence of non-relapse mortality. VII. To assess overall survival and progression-free survival. VIII. To assess the incidence of withdrawal syndrome in patients with myelofibrosis.

TERTIARY OBJECTIVES (CORRELATIVE STUDIES):

I. To study immune recovery and cytokines at various time points pre and post-transplant.

II. To study deoxyribonucleic acid (DNA) damage studies in various cells post-transplant.

OUTLINE:

CONDITIONING CHEMOTHERAPY: Patients receive busulfan intravenously (IV) over 3 hours on days -20, -13, and -6 to -3, and fludarabine IV over 1 hour on days -6 to -3 in the absence of disease progression or unacceptable toxicity.

ALLOGENEIC STEM CELL TRANSPLANTATION: Patients undergo ASCT on day 0.

GVHD PROPHYLAXIS: Patients receive itacitinib orally (PO) once daily (QD) on days -21 to 80. Patients with no evidence of GVHD at day 80 receive a tapered dose of itacitinib until day 90. Patients also receive tacrolimus IV then PO twice daily (BID) for 3 months when able, and methotrexate IV over 30 minutes on days 1, 3, and 6 (day 11 also for patients with a matched unrelated donor).

After completion of study treatment, patients are followed up at 100 days, 6 months, and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky performance status of at least 70
* Patients with hematological disorders undergoing ASCT with conditioning regimen of timed sequential busulfan and fludarabine
* Human leukocyte antigen (HLA)-identical sibling or 8/8 matched unrelated donor available
* Life expectancy of at least 12 weeks (3 months)
* Direct bilirubin not greater than 1 mg/dL
* Alanine transaminase (ALT) less than or equal 3 x upper limit of normal range
* Serum creatinine less than 1.5 x the upper limit of normal range and creatinine clearance greater than 50 ml/min
* Diffusing capacity for carbon monoxide (DLCO) 65% of predicted corrected for hemoglobin
* Left ventricle ejection fraction (LVEF) of at least 50%
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of study drug. Post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test
* Subjects (men and women) of childbearing potential must agree to use adequate contraception beginning at the signing of the informed consent until at least 30 days after the last dose of study drug. The definition of adequate contraception will be based on the judgment of the principal investigator or a designated associate

Exclusion Criteria:

* Patients with a comorbidity score > 3. The principal investigator is the final arbiter of eligibility and enrollment of patients with comorbidity score > 3 and may permit enrollment of these patients on individual basis

  * Active or clinically significant cardiac disease including:

    * Congestive heart failure New York Heart Association (NYHA) > class II
    * Active coronary artery disease
    * Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin
    * Unstable angina (anginal symptoms at rest), new-onset angina within 3 months before transplant, or myocardial infarction within 6 months before transplant
* Patients with uncontrolled infections
* Patients with active hepatitis B and C

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Graft versus host disease (GVHD)-free/relapse free survival rate | At 1 year
  The proportion of patients who are alive without disease relapse of GVHD at one year will be reported, along with the corresponding 95% confidence interval. Logistic regression will be used to assess the association between success and clinical and treatment covariates of interest.

SECONDARY OUTCOMES:
Time to neutrophil engraftment | Up to day 42
  Will be calculated from the time of transplant and estimated by the Kaplan-Meier method. Distributions will be compared between patients with matched and mismatched donors via the long-rank test.
Time to platelet engraftment | Up to day 42
  Will be calculated from the time of transplant and estimated by the Kaplan-Meier method. Distributions will be compared between patients with matched and mismatched donors via the long-rank test.
To assess the incidence of non-relapse mortality | At day 100
To assess the toxicity profile associated with this regimen | Up to 1 year
To assess the incidence of acute and chronic GVHD. | Up to 1 year
Time to disease relapse | Up to 1 year
  Will be modeled using Cox proportional hazards regression models, considering clinical, demographic, and treatment covariates of interest.
Incidence of non-relapse mortality | Up to 1 year
  Will be modeled using Cox proportional hazards regression models, considering clinical, demographic, and treatment covariates of interest. Will be assessed in a competing risks framework, with similar analyses performed.
To assess overall survival and progression-free survival. | From day of transplant until day of death, assessed up to 1 year
Incidence of withdrawal syndrome in patients with myelofibrosis | Up to 1 year

OTHER OUTCOMES:
Immune recovery and cytokines | Up to 1 year
  Generalized linear mixed models will be used to assess the association between cytokines over time and treatment and other factors.
Deoxyribonucleic acid (DNA) damage studies | Up to 1 year
  The proportion of patients with DNA damage will be reported, and generalized logistic mixed models may be used to assess the association with similar covariates.

CONTACTS AND LOCATIONS:
Overall Officials: Uday R Popat, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States